CLINICAL TRIAL: NCT04053790
Title: Evaluation of the Effectiveness and Safety of Lactobacillus Fermentum and Lactobacillus Delbrueckii (Lactobacillus LB) in the Treatment of Patients With Irritable Bowel Syndrome With Predominance of Diarrhea (IBS-D)
Brief Title: Lactobacillus LB as Treatment for Irritable Bowel Syndrome With Predominance of Diarrhea (IBS-D)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, MARIA DE FATIMA HIGUERA DE LA TIJERA, Head of Gastroenterology and Hepatology Department, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DI/18/107/03/080
Record Dates: First submitted 2019-02-20; First posted 2019-08-13 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: irritable bowel syndrome with diarrhea; Lactobacillus LB; treatment; safety; efficacy
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo group (Placebo Comparator): Patients in this group will receive placebo 1 tablet every 12 hours, during 4 weeks.
  Interventions: Other: placebo
- LB 10000 (Active Comparator): Patients in this group will receive placebo 1 tablet containing 5,000 millions of lactobacillus LB, every 12 hours, during 4 weeks.
  Interventions: Drug: lactobacillus LB
- LB 20000 (Active Comparator): Patients in this group will receive placebo 1 tablet containing 10,000 millions of lactobacillus LB, every 12 hours, during 4 weeks.
  Interventions: Drug: lactobacillus LB

INTERVENTIONS:
Drug: lactobacillus LB — administration of different doses of Lactobacillus LB according to the treatment groups described previously
  Other Names: Lactobacillus fermentum + lactobacillus delbrueckii, lyophilized powder; Lacteol
  Arms: LB 10000; LB 20000
Other: placebo — a tablet of placebo every 12 hours given by mouth
  Other Names: inactive principle
  Arms: placebo group

SUMMARY:
Background: The combination of Lactobacillus fermentum and Lactobacillus delbrueckii (Lactobacillus LB) has proven to be effective and safe for the treatment of acute diarrhea in children. Also, a clinical trial in adult patients with chronic diarrhea, showed a reduction in the number of daily stools. However, the evidence is not enough regarding the efficacy and safety of Lactobacillus LB for treatment of patients with irritable bowel syndrome with predominance of diarrhea (IBS-D).

Justification for this study: Lactobacillus LB could be a promising treatment for patients with IBS-D; nevertheless, the scientific evidence in this context is limited and it is not recent. Therefore, is necessary to explore the efficacy and safety of Lactobacillus LB in patients with IBS-D according to Rome IV criteria.

Hypothesis: Lactobacillus LB is useful to decrease the frequency and improve the stools consistency of patients diagnosed with IBS-D by Rome IV criteria.

Primary Outcome: To compare the treatment with Lactobacillus LB at two different doses: a) 20,000 million / day, vs. b) 10,000 million / day; and to determine if one of them is better than c) placebo, to decrease the frequency (weekly average of the number of stools/day) in patients diagnosed with IBS-D by Rome IV criteria.

Design of the study: Clinical trial, randomized, double-blind, placebo-controlled.

Keywords: irritable bowel syndrome with diarrhea, Lactobacillus LB, treatment, efficacy, safety.

DETAILED DESCRIPTION:
Background: The combination of Lactobacillus fermentum and Lactobacillus delbrueckii (Lactobacillus LB) has proven to be effective and safe for the treatment of acute diarrhea in children. Also, a clinical trial in adult patients with chronic diarrhea showed a reduction in the number of daily stools. However, the evidence is not enough regarding the efficacy and safety of Lactobacillus LB for the treatment of patients with irritable bowel syndrome with a predominance of diarrhea (IBS-D).

Justification for this study: Lactobacillus LB could be a promising treatment for patients with IBS-D; nevertheless, the scientific evidence in this context is limited and it is not recent. Therefore, is necessary to explore the efficacy and safety of Lactobacillus LB in patients with IBS-D according to Rome IV criteria.

Hypothesis: Lactobacillus LB is useful to decrease the frequency and improve the stools consistency of patients diagnosed with IBS-D by Rome IV criteria.

Primary Outcome: To compare the treatment with Lactobacillus LB at two different doses: a) 20,000 million / day, vs. b) 10,000 million / day; and to determine if one of them is better than c) placebo, to decrease the frequency (weekly average of the number of stools/day) in patients diagnosed with IBS-D by Rome IV criteria.

Design of the study: Clinical trial, randomized, double-blind, placebo-controlled.

Keywords: irritable bowel syndrome with diarrhea, Lactobacillus LB, treatment, efficacy, safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting Rome IV criteria for IBS-D, without specific medical treatment for the last 4 weeks prior to inclusion in this study.

Exclusion Criteria:

* Presence of any chronic organic disease, consumption of any medication, patients with alterations in blood cell count, erythrocyte sedimentation rate, thyroid function tests, liver function tests, blood chemistry, anti-endomysial or anti-transglutaminase antibodies, positive test for presence of blood in stools, fecal calprotectin > 50mcg/g. Also, those who do not sign informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2023-01-29 (Actual)

PRIMARY OUTCOMES:
decrease in the number of stools per day | 4 weeks
  weekly average number of evacuations / day, comparing before and after treatment

SECONDARY OUTCOMES:
improvement in the consistency of the stools according to Bristol scale. | 4 weeks
  Bristol scale: type 1= separate hard lumps, type 2= sausage shaped but lumpy, type 3= like a sausage but with cracks on ots surface, type 4= like a sausage or sanake, smooth and soft, type 5= soft blobs with clear cut-edges, type 6= fluffy pieces with ragged edges, a mushy stool, type 7 = watery, no solid pieces.
improvement in bloating measured by a Likert scale (0-4) | 4 weeks
  Likert scale: 0=without bloating, 1=mild bloating, 2=moderate bloating, 3=severe bloating
improvement in abdominal pain measured by a Likert scale (0-4) | 4 weeks
  Likert scale: 0=without pain, 1=mild pain, 2=moderate pain, 3=severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Higuera de la Tijera, MD, PhD, Principal Investigator — Hospital General de Mexico
Locations (1):
- Hospital General de Mexico, Mexico City, Choose Any State/Province, Mexico